CLINICAL TRIAL: NCT01184365
Title: Spinal Cord Injury Energy Management Program
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H10-01037; NSP-104021 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2010-08-11; First posted 2010-08-18 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Spinal Cord Injury
Keywords: fatigue; energy management; spinal cord injury; self-efficacy; environment
MeSH Terms: conditions — Spinal Cord Injuries; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EnMP-1 (Experimental): The goal of the EnMP-1 is to enable participants, through a behavioural, psycho-educational intervention, to better manage and understand their fatigue. This program is provided in four, two-hour sessions held weekly.
  Interventions: Behavioral: Energy Management Program
- EnMP-2 (Active Comparator): The goal of the EnMP-2 is to control for group effects
  Interventions: Behavioral: Energy Management Program

INTERVENTIONS:
Behavioral: Energy Management Program — The program content over the four sessions is structured as follows: Session 1 is an introduction to the group, important concepts, and upcoming session topics; Session 2 further elaborates on the concepts introduced in session 1 and encourages self-reflection; Session 3 is the peer to peer contact by phone or in person to assist with problems and share tips that really worked; and Session 4 concludes the program and serves to consolidate information learned.
  Arms: EnMP-1
Behavioral: Energy Management Program — The goal of the EnMP-2 is to control for group effects
  Arms: EnMP-2

SUMMARY:
Fatigue is a common complaint of persons with spinal cord injury (SCI) that negatively affects physical function, participation in daily activities, employment, and community involvement. No behavioural intervention for fatigue has been reported for SCI, though the benefits of such programs have been proven in persons with neurological conditions like multiple sclerosis and arthritis. Based on a study with people with SCI, an energy management program (EnMP-1) was developed. The focus of this study is to test EnMP-1. Adults with SCI living in the community and reporting fatigue as a problem will participate in the program.

Hypothesis: Participants in the EnMP-1 group will show significantly lower fatigue impact scores and higher self-efficacy scores immediately after, 3 months, and 6 months post-intervention than EnMP-2 participants.

DETAILED DESCRIPTION:
Detailed Description Extended description of the protocol (Background, purpose, hypothesis, and inclusion/exclusion criteria already contained in other fields):

The protocol subjects will follow is conceptualized into three periods: the pre-program phase, the program phase of either the EnMP-1 or the EnMP-2, and the follow-up phase.

Pre-program Phase: Potential subjects will contact the Research Coordinator to volunteer for the study and to have any questions addressed. At that time, subjects will be screened by phone or in person using a Participant Screening Questionnaire to ensure that they meet the inclusion/exclusion criteria of the study. If the individual is deemed eligible, the Research Coordinator will gather demographic information and provide or forward the participant the pre-program preparation package that includes: a fact sheet about the study; the consent form; self-reported study measures (one primary for fatigue, one secondary for self-efficacy, and four co-variate measures assessing depression, pain, and sleep); and a self-addressed, stamped return envelope. Participants will be contacted one week after the pre-program package has been sent, to address questions and to verbally assist in completing the outcome measures, if required. They will be asked to sign the consent form, complete the study measures and return these in the envelope provided in the package.

Four weeks later (one-week before the program phase) subjects will be forwarded the study measures to complete prior to the first session. Subjects will be contacted 1-2 days before the first session to address concerns, clarify that measures are to be completed and brought to the first session, and to remind subjects of the date, time and location of the first session. Subjects who received the workbook will be encouraged to browse and review its content. The study measures will be collected at the beginning of the first session.

Program Phase: All subjects will participate in the four, two-hour sessions held one week apart for four weeks.

The program content for both the EnMP-1 and EnMp-2 group sessions is structured as follows: Session 1 is an introduction to the group, important concepts, and upcoming session topics; Session 2 further elaborates on the concepts introduced in session 1 and encourages self-reflection; Session 3 is the peer to peer contact by phone or in person to assist with problems and share tips that really worked; and Session 4 concludes the program and serves to consolidate information learned.

At the conclusion of the week-four session, subjects will be provided with a package that includes the study measures, a program evaluation and self-addressed stamped envelope. They will be asked to complete the measures and the evaluation over next week and return them in the envelope provided. Subjects will be contacted 1-2 days after this last session to address questions and to remind them to return the measures and program evaluation in the envelope provided. After one-week, if the package has not been received, subjects will be contacted to assist with any issues and to encourage return of the package. This will be repeated one further time to maximize return.

Follow-up Phase: After the program phase is concluded, there will be a six-month follow-up. Subjects will be forwarded the self-report study measures and self-addressed stamped envelope and asked to complete and return them in the envelope provided. Subjects will be contacted one week after the package is sent to address questions and to remind them to return the measures in the envelope provided. If the package has not been received, after another week, subjects will be contacted to assist with any issues and to encourage return of the package. This will be repeated one further time, a week later, to maximize return.

The time commitment for participating in this study is between 11-12 hours over 7 months.

ELIGIBILITY:
Inclusion Criteria:

* must reside in the community in the Lower Mainland of Vancouver, British Columbia, Canada
* must be an adult (19-65 years old)
* be English speaking
* have a spinal cord injury and is living in the community
* experiencing problems with managing energy that may or may not result in difficulty participating at home, work or in the community.

Exclusion Criteria:

* have a severe brain injury that may prevent their participation in the study
* have other conditions such as arthritis, multiple sclerosis, cancer, or anemia

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To test a behavioural (not pharmaceutical or surgical) intervention for fatigue in SCI | Six months
  The primary outcome measure evaluates fatigue impact and is the Modified Fatigue Impact Scale (MFIS-SCI) which was originally developed for individuals with MS and was modified and tested by members of the research team in a study of fatigue in a sub-acute sample of individuals with SCI.

SECONDARY OUTCOMES:
Evaluates self-efficacy and is the Self-Efficacy for Performing Energy Conservation Strategies Assessment (SEPECSA) | Six months
  The measure consists of items regarding confidence in employing various means of energy conservation and is answered on a scale of 1-10, with one being not at all confident to ten being completely confident.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Forwell, PhD, OT(C), FCAOT, Principal Investigator — University of British Columbia; William C. Miller, Dr., Study Director — University of British Columbia; Andrea Townson, Dr., Study Director — University of British Columbia; Karen Hammell, Dr., Study Director — University of British Columbia
Locations (1):
- Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada